CLINICAL TRIAL: NCT01050530
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial to Investigate the Efficacy of OPC-41061 Administered at a Dose of 7.5 mg in Patients With Hepatic Edema
Brief Title: A Trial to Investigate the Efficacy of OPC-41061 Administered at a Dose of 7.5 mg in Patients With Hepatic Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-08-001; JapicCTI-100982
Record Dates: First submitted 2010-01-07; First posted 2010-01-15 (Estimated); Results first posted 2014-01-31 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Cirrhosis
Keywords: Cirrhosis; ascites; Tolvaptan; OPC-41061
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPC-41061 (Experimental)
  Interventions: Drug: OPC-41061
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC-41061 — Once-daily oral administration of OPC-41061 at 7.5 mg after breakfast for 7 days
  Arms: OPC-41061
Drug: Placebo — Once-daily oral administration of placebo after breakfast for 7 days
  Arms: Placebo

SUMMARY:
OPC-41061 at 7.5 mg/day or placebo will be orally administered once daily for 7 days to cirrhosis patients with ascites despite having received treatment with conventional diuretics and the change in body weight from baseline at the time of the final administration will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients judged as having cirrhosis based on previous imaging diagnosis

  * Definition of cirrhosis includes patients with collateral circulation due to chronic hepatic impairment
* Patients with ascites in whom the dose of existing diuretics cannot be increased due to risk of adverse drug reactions such as electrolyte abnormalities, or in whom sufficient therapeutic effect cannot be obtained with existing diuretics
* Patients who have been receiving oral combination therapy with a loop diuretic and an anti-aldosterone agent from at least 7 days prior to receipt of informed consent, with a dose combination of either loop diuretic equivalent to furosemide 40 mg/day or higher plus spironolactone 25 mg/day or higher, or loop diuretic equivalent to furosemide 20 mg/day or higher plus spironolactone 50 mg/day or higher
* Patients who are hospitalized or who can be hospitalized for the trial
* Patients capable of giving informed consent
* Patients who, together with their partner, agree to use an appropriate method of contraception until 4 weeks after the final trial drug administration

Exclusion Criteria:

* Patients with any of the following complications or symptoms:
* Hepatic encephalopathy (hepatic coma of grade 2 or higher)
* Hepatocellular carcinoma with imaging-diagnosed vascular infiltration into trunk or primary branch of portal vein, inferior vena cava, or trunk of hepatic vein
* Endoscopic findings from screening examination or from within 30 days prior to screening examination indicating the need for new therapy for esophageal or gastric varices during the trial period
* Repeated hemorrhoidal bleeding due to rectal varicose veins within 30 days prior to informed consent
* Heart failure (New York Heart Association Class III or IV)
* Anuria
* Impaired urination due to urinary tract stricture, urinary calculus, tumor in urinary tract, or other cause
* Patients with a history of any of the following disorders:
* Cerebrovascular disorder within 30 days prior to informed consent
* Hypersensitivity or idiosyncratic reaction to benzazepine derivatives (such as mozavaptan hydrochloride or benazepril hydrochloride)
* Morbidly obese patients with a body mass index (BMI: body weight (kg)/height (m)2) exceeding 35
* Patients with sitting systolic blood pressure lower than 90 mmHg
* Patients with any of following abnormal clinical laboratory values at time of the screening examination: Hemoglobin lower than 8.0 g/dL, total bilirubin higher than 4.0 mg/dL, serum creatinine higher than 2.0 mg/dL, serum sodium higher than 147 mEq/L, or serum potassium higher than 5.5 mEq/L
* Patients who are unable to take oral medication
* Female patients who are pregnant, possibly pregnant, or breast-feeding, or who are planning to become pregnant
* Patients who have used albumin preparations (therapeutic agents for hypoalbuminemia) or blood products containing albumin from within 7 days prior to informed consent
* Patients who received any investigational drug other than OPC-41061 within 30 days prior to informed consent
* Patients who have previously received OPC-41061
* Any patient who, in the opinion of the principle investigator or subinvestigator, is inappropriate for participation in the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OPC-41061 | Placebo
Started | 82 | 80
Completed | 74 | 70
Not Completed | 8 | 10
Not completed — Adverse Event | 6 | 3
Not completed — Lack of Efficacy | 1 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-41061 | Placebo | Total
Number analyzed (Participants) | 82 | 80 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.4) | 66.4 (8.7) | 66.4 (9.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 29 | 61
  >=65 years | 50 | 51 | 101
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 61
  Male | 52 | 49 | 101
Region of Enrollment [Number; unit: participants]
  Japan | 82 | 80 | 162

OUTCOME MEASURES:

1. Primary Outcome: Body ｗeight
Description: Change in body weight from baseline after 7-day repeated oral administration of OPC
Time Frame: Baseline, Day 7 or at the discontinued of treatment
Population: Full Analysis Set; LOCF
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | OPC-41061 | Placebo
Number analyzed (Participants) | 82 | 80
Kg | -1.95 (1.77) | -0.44 (1.93)
Statistical Analysis 1: Comparison: OPC-41061 vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -1.51, 95% CI 2-sided [-2.08 to -0.93]

2. Secondary Outcome: Ascites Volume
Description: Change in ascites volume from baseline as measured by CT at end of treatment
Time Frame: Baseline, Day 7 or at the discontinued of treatment
Population: Full Analysis Set; LOCF
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | OPC-41061 | Placebo
Number analyzed (Participants) | 82 | 80
mL | -492.4 (760.3) | -191.8 (690.8)
Statistical Analysis 1: Comparison: OPC-41061 vs Placebo; Test type: Superiority or Other; p = 0.0093, t-test, 2 sided; Mean Difference (Final Values) = -300.7, 95% CI 2-sided [-526.2 to -75.1]

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | OPC-41061 | Placebo
Serious Adverse Events (participants affected / at risk) | 7/82 | 10/80
Other Adverse Events (participants affected / at risk) | 36/82 | 26/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPC-41061 (N=82) | Placebo (N=80)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pylethrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Omphalitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Coma Hepatic (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 1 (1) | 3 (3)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Respiration Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intra-Abdominal Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPC-41061 (N=82) | Placebo (N=80)
Constipation (Gastrointestinal disorders) | 6 (6) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (5) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Thirst (General disorders) | 11 (12) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 6 (7)
Blood Urea Increased (Investigations) | 1 (1) | 4 (4)
Hyperammonaemia (Investigations) | 2 (2) | 3 (3)
Hepatic Encephalopathy (Nervous system disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 6 (6) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 5 (5) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No